CLINICAL TRIAL: NCT05991336
Title: Growth and Development, Health-related Quality of Life of Children With Transfusion-dependent Beta-thalassemia After Gene Therapy
Brief Title: Growth and Development-related Outcomes in Children With Transfusion-dependent Beta-thalassemia After Gene Therapy
Status: Recruiting | Type: Observational
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Principal Investigator, Jun Shi, Director, Regenerative Medicine Clinic Center, Institute of Hematology & Blood Diseases Hospital, China
Other Study IDs: GDH-001
Record Dates: First submitted 2023-07-27; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Transfusion-dependent Beta-Thalassemia; Gene Therapy
Keywords: Transfusion-dependent Beta-Thalassemia; gene therapy; cohort study; case-control
MeSH Terms: interventions — Genetic Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The peripheral blood sample was collected and stored in the IHBDH biobank.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Gene therapy group: TDT Children who have received gene therapy between 3~14 years old.
  Interventions: Genetic: Gene therapy
- Supportive therapy group: TDT Children who received lifelong treatment with blood transfusions and iron chelation. They were selected based on the age and sex of the gene therapy group.
- Healthy children group: Healthy children were selected based on the age and sex of the gene therapy group.

INTERVENTIONS:
Genetic: Gene therapy — Autologous edited hematopoietic stem cell transplantation
  Groups: Gene therapy group

SUMMARY:
The investigate will conduct a cohort study to compare the growth and development, metabolism, lifestyle behavior, and health-related quality of life among three groups: children with transfusion-dependent β-thalassemia (TDT) who have received gene therapy, TDT children with lifelong supportive therapy and healthy children.

ELIGIBILITY:
Inclusion Criteria:

Gene therapy group-inclusion

* Male or female age of 3-14 years
* TDT Children who have received gene therapy.
* Subjects who are willing and able to provide written informed consent.

Supportive therapy group-inclusion

* Gender same as the matched case
* Age similar to the matched case
* Children with β-TDT
* No history of gene therapy or allogeneic hematopoietic stem cell transplantation
* Subjects who are willing and able to provide written informed consent.

Healthy children group-inclusion

* Gender same as the matched case
* Age similar to the matched case
* Subjects who are willing and able to provide written informed consent.

Exclusion Criteria:

* Diagnosis of compound α-thalassemia
* Uncontrolled systemic fungal, bacterial, or viral infection
* History of malignant solid tumors, myeloproliferative or immunodeficiency diseases
* Diagnosed with mental illness
* Patients considered to be ineligible for the study by the investigator for reasons other than the above

Discontinuation of Study :

* Subjects who are unwilling or unable to continue participating in the study (withdrawal of informed consent) may withdraw from the study
* Subjects who received gene therapy or allogeneic hematopoietic stem cell transplantation during the study
* The subject is seriously non-compliant with the study requirements, such as missing 2 consecutive visits
* Subject lost to follow-up

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants are divided into three groups: TDT children who have received gene therapy, TDT children who have received lifelong supportive therapy, and healthy children.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-06-05 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Growth in pediatric subjects will be assessed by height. | Up to 5 years.
  Height in meters.
Growth in pediatric subjects will be assessed by weight. | Up to 5 years.
  Weight in kilograms.
Growth in pediatric subjects will be assessed by the head and chest circumference. | Up to 5 years.
  Head and chest circumference in centimeters.
Growth in pediatric subjects will be assessed by interocular distance. | Up to 5 years.
  Interocular distance in centimeters.
Growth in pediatric subjects will be assessed by bone density. | Up to 5 years.
  Bone density measurement is measured by a procedure called densitometry, performed in the radiology medicine departments of hospitals or clinics. The result is the bone mineral density in grams per unit area (g/cm2).
The pubertal status will be measured using by Tanner scale. | Up to 5 years.
  The Tanner scale, a well-known technique used to define pubertal stage, is based on physical measurements of development based on external primary and secondary sex characteristics (from Tanner 1: pre-pubertal to Tanner 5: mature adolescent).It was developed by Marshall and Tanner while conducting a longitudinal study during the 1940s to the 1960s in England. Based on observational data, they developed separate scales for the development of external genitalia: phallus, scrotum, and testes volume in males; breasts in females; and pubic hair in both males and females.
Hormonal levels will be measured by clinical examination. | Up to 5 years.
  Hormonal levels included thyroid-stimulating hormone (TSH), serum triiodothyronine (T3), serum-free triiodothyronine (T4), growth hormone (GH, including IGF-1 and IGF-2), and sex hormone examination. Sex hormone examination is only for the following subjects: estradiol, FSH and LH for girls aged 9-18; testosterone, FSH and LH for boys aged 12-18.
Quality of life will be measured using by Pediatric Quality of Life Inventory (PedsQL) at baseline and the end of the study. | Up to 5 years.
  The Pediatric Quality of Life Inventory (PedsQL) is a valid, standardized, generic, and self-reporting assessment tool to measure health-related quality of life HRQOL for pediatrics and adolescents. PedsQL contain 23-items, and consists of the following: physical functioning, emotional functioning, social functioning, and school functioning. Each item is scored on a 5-point scale, scores are linearly transformed to a 0-100 scale in which high score means better condition.
Lifestyle behaviors will be assessed by general questioning. | Up to 5 years.

CONTACTS AND LOCATIONS:
Locations (1):
- Regenerative Medicine Center, Tianjin, Tianjin Municipality, China